CLINICAL TRIAL: NCT06100471
Title: Evaluation of Genetic Signature in Endometriosis Disease by Non Invasive Sampling
Acronym: niEndometriosi
Status: Enrolling by invitation | Type: Observational
Sponsor: Eurofins Genoma (Industry)
Responsible Party: Sponsor
Other Study IDs: 01-23
Record Dates: First submitted 2023-10-13; First posted 2023-10-25 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Endometriosis; Hypofertility
Keywords: endo
MeSH Terms: conditions — Endometriosis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — tissue biopsy and saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- case: Patients with endometriotic adnexal pathology
  Interventions: Other: Observational study
- control: Patients with non endometriotic adnexal pathology
  Interventions: Other: Observational study
- analytical control: Patients with no gynecological pathology, not undergoing surgery
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study in different tissues in identifing new genetic markers related to endometriosis disease

SUMMARY:
Endometriosis is a disease that affects 10-15% of the general population and 50% of infertile women. It is characterized by the presence of endometrial tissue outside the uterine cavity. Endometriosis can lead to infertility by interfering through endocrine and mechanical alterations on the function of the ovaries, fallopian tubes, and uterus. The aim of the study is to define the differential expression of a cluster of RNAs tissue driven for the identification of an RNA profile in saliva, specific for endometriosis. This study focuses on the expression of genes involved in the control and regulation of apoptosis, cell survival, metabolism, cell adhesion and invasion, angiogenesis, inflammation, and estrogen receptor expression levels.

DETAILED DESCRIPTION:
Retrospective selection based on anamnestic criteria of: 50 patients with diagnosed endometriotic adnexal pathology (case, CA), 50 patients with non-endometriotic adnexal pathology (control, CO) and 50 patients with no gynecological pathology, not undergoing surgery (analytical control).

The study involves collecting a saliva sample from all patients involved in the study, and performing a biopsy from both patients with endometriotic adnexal pathology (CA) and patients with non-endometriotic adnexal pathology (CO).

ELIGIBILITY:
Inclusion Criteria:

* Case population (CA), patients with endometriotic adnexal pathology
* Control population (CO), patients with non-endometriotic adnexal pathology
* Analytical control population (C-), patients with no gynecologic pathology, not undergoing surgery

Exclusion Criteria:

* Women with ages outside the inclusion range
* Pregnant patient
* Patient with a personal history of cancer
* Patient infected with HIV

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Groups of study:
  * patients with diagnosed endometriotic adnexal pathology (case, CA)
  * patients with non-endometriotic adnexal pathology (control, CO)
  * patients with no gynecological pathology, not undergoing surgery (analytical control)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Next Generation Sequencing technical validation | 1 month
  Assessing the quality of Next Generation Sequencing via the FASTQC tool. Following benchmarks will be considered:
  1.1 Per base sequence quality [Phred score: positive real number, the higher the better] 1.2 Total number of sequenced reads [integer: positiver integer number, the higher the better]
Wet lab kit validation | 1 month
  Assessing the quality of the kit by mapping the reads against public miRNA databases. Following benchmark will be considered: Total reads mapped [integer]

SECONDARY OUTCOMES:
Tissue validation | 2 months
  Genetic profiling of miRNOME from saliva versus FFPE-tissues
Clinical validation | 4 months
  Correlation of miRNOME signature in saliva among cases, controls and analytical groups
Biomarkers identification | 7 months
  Identification of specific signature related to endometriosis, with at least 2 Log2fold change

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Genoma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dabi Y, Suisse S, Puchar A, Delbos L, Poilblanc M, Descamps P, Haury J, Golfier F, Jornea L, Bouteiller D, Touboul C, Darai E, Bendifallah S. Endometriosis-associated infertility diagnosis based on saliva microRNA signatures. Reprod Biomed Online. 2023 Jan;46(1):138-149. doi: 10.1016/j.rbmo.2022.09.019. Epub 2022 Sep 27. PMID 36411203
- [Background] Bendifallah S, Dabi Y, Suisse S, Jornea L, Bouteiller D, Touboul C, Puchar A, Darai E. A Bioinformatics Approach to MicroRNA-Sequencing Analysis Based on Human Saliva Samples of Patients with Endometriosis. Int J Mol Sci. 2022 Jul 21;23(14):8045. doi: 10.3390/ijms23148045. PMID 35887388
- [Background] Bendifallah S, Suisse S, Puchar A, Delbos L, Poilblanc M, Descamps P, Golfier F, Jornea L, Bouteiller D, Touboul C, Dabi Y, Darai E. Salivary MicroRNA Signature for Diagnosis of Endometriosis. J Clin Med. 2022 Jan 26;11(3):612. doi: 10.3390/jcm11030612. PMID 35160066
- [Background] Bendifallah S, Dabi Y, Suisse S, Jornea L, Bouteiller D, Touboul C, Puchar A, Darai E. MicroRNome analysis generates a blood-based signature for endometriosis. Sci Rep. 2022 Mar 8;12(1):4051. doi: 10.1038/s41598-022-07771-7. PMID 35260677
- [Background] Dabi Y, Suisse S, Jornea L, Bouteiller D, Touboul C, Puchar A, Darai E, Bendifallah S. Clues for Improving the Pathophysiology Knowledge for Endometriosis Using Plasma Micro-RNA Expression. Diagnostics (Basel). 2022 Jan 12;12(1):175. doi: 10.3390/diagnostics12010175. PMID 35054341
- [Background] Bendifallah S, Puchar A, Suisse S, Delbos L, Poilblanc M, Descamps P, Golfier F, Touboul C, Dabi Y, Darai E. Machine learning algorithms as new screening approach for patients with endometriosis. Sci Rep. 2022 Jan 12;12(1):639. doi: 10.1038/s41598-021-04637-2. PMID 35022502